CLINICAL TRIAL: NCT03457753
Title: A Multi-Center, Open Label Study to Assess the Safety and Tolerability of Riluzole Oral Soluble Film in Subjects With Amyotrophic Lateral Sclerosis Over 12 Weeks of Twice Daily Treatment.
Brief Title: Riluzole Oral Soluble Film Safety and Tolerability in Amyotrophic Lateral Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor stopped the study due to a change in study plans
Sponsor: Aquestive Therapeutics (Industry)
Collaborators: Inventiv Health (Unknown); Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17MO1R-0016
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: ALS
Keywords: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open label safety and tolerability trial. Approximately twenty-five (25) individuals with amyotrophic lateral sclerosis (ALS) will be enrolled.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with ALS (Experimental): Riluzole Oral Soluble Film (ROSF) 50 mg will be administered in subjects with ALS twice daily. It is intended that at least five (5) of the twenty-five (25) subjects enrolled will be subjects scoring greater than 20 on the Eating Assessment Tool (EAT-10) (representative of ALS patients reporting moderate swallowing impairments in a patient report validated scale).
  Interventions: Drug: Riluzole Oral Soluble Film

INTERVENTIONS:
Drug: Riluzole Oral Soluble Film — Riluzole Oral Soluble Film (ROSF) containing Riluzole 50mg .
  Other Names: ROSF

SUMMARY:
The primary objective of this study is to assess the safety and tolerability, with emphasis on the oral cavity, of ROSF (containing riluzole 50mg) in subjects with amyotrophic lateral sclerosis (ALS) administered twice daily for 12 weeks. Secondary objectives include (1) to record the subject's assessment of any difficulty taking riluzole administered as ROSF and any difficulty taking riluzole in the tablet formulation and (2) to record the relative preference, if any, of subjects and caretakers, for riluzole administered as ROSF vs. the riluzole tablet.

DETAILED DESCRIPTION:
The total study participant time is expected to be approximately 14 weeks from time of screening to completion of study. Subjects will be instructed on the use of ROSF and receive the first dose of ROSF under supervision of the investigator during Visit 1.Subjects will then continue on ROSF 50mg twice daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, between 18-80 years of age, inclusive.
2. Subjects having a diagnosis of probable or definite ALS in accordance with the Revisited El-Escorial Criteria.
3. Subjects must have no known allergy to riluzole or inactive ingredients* in ROSF.
4. Subjects or subject's legally authorized representative must be willing and able to complete informed consent/assent and HIPAA authorization.
5. Ability to comprehend and be informed of the nature of the study, as assessed by the Primary or Sub-Investigator.
6. Subjects prescribed to take riluzole at or before the time of first dose. (The study is open to subjects currently taking riluzole at screening, subjects who are not currently taking riluzole at screening but who have taken riluzole in the past, and subjects to be newly started on riluzole (given as ROSF in the course of this study).
7. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
8. Female subjects of childbearing potential must have a negative urine pregnancy test at Screening and Visit 1-3. Female subjects of childbearing potential (i.e. not surgically sterile, not 2 years postmenopausal, or not with a sterile partner) must have a negative pregnancy test at screening and Visit 1-3, agree to abstinence, practicing double barrier contraception or using an FDA approved barrier method contraceptive (e.g., licensed hormonal or barrier methods) for greater than 2 months prior to screening visit and commit to an acceptable form of birth control for the duration of the study and for 30 days after participation in the study.
9. Subjects, in the judgment of the investigator, must be suitable candidates for administration of ROSF (riluzole oral soluble film).

Exclusion Criteria:

1. Subjects with a history of clinically significant liver disease, renal disease, or any other medical condition judged to be exclusionary by the investigator.
2. Subjects who are unwilling to sign informed consent or subjects who for any other reason in the judgment of investigator are unable to complete the study.
3. Female subjects who have a positive urine pregnancy test (βhCG) at screening or visit 1, are trying to become pregnant or are breastfeeding.
4. Subjects with active cancer within the previous 2 years, except treated basal cell carcinoma of the skin.
5. Subjects who have taken any experimental drug within 30 days prior to enrollment or within 5 half-lives of the investigational drug -whichever is the longer period. However, subjects who have previously completed other Aquestive sponsored ROSF clinical studies within the last 30 days prior to enrollment may be eligible for consideration for entry into this study.
6. Subjects with known history or presence of moderate or severe renal impairment as defined by a calculated creatinine clearance of ≤50 mL/minute.
7. Subjects currently taking riluzole with alanine aminotransferase (ALT) levels greater than 5 times upper limit of normal or with evidence of clinical jaundice. (Riluzole should be discontinued in these patients.)
8. Subjects who will be receiving riluzole for the first time who exhibit baseline elevations of several liver function tests (especially elevated bilirubin). (These findings at baseline should preclude the use of riluzole including ROSF.)
9. Use of potentially hepatotoxic drugs: (e.g., allopurinol, methyldopa, sulfasalazine).
10. Subjects with clinically significant abnormal laboratory values in the judgment of the investigator.
11. Use of strong or moderate CYP1A2 inhibitors (e.g., ciprofloxacin, enoxacin, fluvoxamine, methoxsalen, mexiletine, thiabendazole, vemurafenib, zileuton) and CYP1A2 inducers (e.g. rifampin and barbiturates) in the previous 30 days before first drug administration.
12. Employee or immediate relative of an employee of the investigator, MonoSol Rx LLC, any of its affiliates or partners, or inVentiv Health.
13. Anything else that, in the opinion of the investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in NCI-CTC score at week 12 | Week 12 (visit 3)
  The National Cancer Institute Common Toxicity Criteria (NCI-CTC) score will be used to evaluate the presence or level of oral cavity irritation on an oral examination, with a grading scale ranging from Grade 0 -5 (0 = no toxicity, 1 = painless ulcers, erythema, or mild soreness, 2 = painful erythema, edema, or ulcers but eating or swallowing possible, 3 = painful erythema, edema, or ulcers requiring intravenous hydration, 4 = severe ulceration, and 5 = death related to toxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Plowman, PhD, CCC-SLP, Principal Investigator — University of Florida; James Wymer, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- Texas Neurology, P.A., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No